CLINICAL TRIAL: NCT02009449
Title: A Phase 1, Open-Label Dose Escalation First-in-Human Study to Evaluate the Tolerability, Safety, Maximum Tolerated Dose, Preliminary Clinical Activity and Pharmacokinetics of AM0010 in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of Pegilodecakin (LY3500518) in Participants With Advanced Solid Tumors
Acronym: IVY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ARMO BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17159; J1L-AM-JZGA (Other: Eli Lilly and Company); AM0010-001 (Other: ARMO BioSciences)
Record Dates: First submitted 2013-12-02; First posted 2013-12-12 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Melanoma; Prostate Cancer; Ovarian Cancer; Renal Cell Carcinoma; Colorectal Carcinoma; Pancreatic Carcinoma; Non-small Cell Lung Carcinoma; Solid Tumors; Breast Cancer
Keywords: Phase 1/Phase 1b; Oncology; Cancer; Solid Tumors
MeSH Terms: conditions — Melanoma; Prostatic Neoplasms; Ovarian Neoplasms; Carcinoma, Renal Cell; Colorectal Neoplasms; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Neoplasms | interventions — pegilodecakin; AM0010; Paclitaxel; Docetaxel; Carboplatin; Cisplatin; Folfox protocol; Oxaliplatin; Gemcitabine; Capecitabine; pazopanib; pembrolizumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (24):
- Part A: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (1 ug/kg) - Daily subcutaneous (SC) injections of pegilodecakin for up to 22 months
  Interventions: Drug: Pegilodecakin
- Part A: Dose Escalation Cohort 2 (Experimental): Pegilodecakin (2.5 ug/kg) - Daily subcutaneous injections of pegilodecakin for up to 22 months
  Interventions: Drug: Pegilodecakin
- Part A: Dose Escalation Cohort 3 (Experimental): Pegilodecakin (5 ug/kg) - Daily subcutaneous injections of pegilodecakin for up to 22 months
  Interventions: Drug: Pegilodecakin
- Part A: Dose Escalation Cohort 4 (Experimental): Pegilodecakin (10 ug/kg) - Daily subcutaneous injections of pegilodecakin for up to 22 months
  Interventions: Drug: Pegilodecakin
- Part A: Dose Escalation Cohort 5 (Experimental): Pegilodecakin (20 ug/kg) - Daily subcutaneous injections of pegilodecakin for up to 22 months
  Interventions: Drug: Pegilodecakin
- Part A: Dose Escalation Cohort 6 (Experimental): Pegilodecakin (40 ug/kg) - Daily subcutaneous injections of pegilodecakin for up to 22 months
  Interventions: Drug: Pegilodecakin
- Part A: Dose Expansion Cohort 1 (Experimental): at least 15 RCC participants will be dosed with pegilodecakin for up to 22 months
  Interventions: Drug: Pegilodecakin
- Part B: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (2.5 ug/kg) daily subcutaneous injections with Platinum / Taxane combination Every 21 days, (21 days = 1 cycle) for 5 cycles.
  Day 1
  * Paclitaxel 200/175 mg/m2 IV, or
  * Docetaxel 75/65 mg/m2 IV And
  * Carboplatin AUC 6/5/4 (max. 6x 150mg) IV or
  * Cisplatin 75mg/m2 IV
  Interventions: Drug: Pegilodecakin; Drug: Paclitaxel or Docetaxel and Carboplatin or Cisplatin
- Part B: Dose Escalation Cohort 2 (Experimental): Pegilodecakin (5 ug/kg) daily subcutaneous injections with Platinum / Taxane combination Every 21 days, (21 days = 1 cycle) for 5 cycles.
  Day 1
  * Paclitaxel 200/175 mg/m2 IV, or
  * Docetaxel 75/65 mg/m2 IV And
  * Carboplatin AUC 6/5/4 (max. 6x 150mg) IV or
  * Cisplatin 75mg/m2 IV
  Interventions: Drug: Pegilodecakin; Drug: Paclitaxel or Docetaxel and Carboplatin or Cisplatin
- Part B: Dose Escalation Cohort 3 (Experimental): Pegilodecakin (10 ug/kg) daily subcutaneous injections with Platinum / Taxane combination Every 21 days, (21 days = 1 cycle) for 5 cycles.
  Day 1
  * Paclitaxel 200/175 mg/m2 IV, or
  * Docetaxel 75/65 mg/m2 IV And
  * Carboplatin AUC 6/5/4 (max. 6x 150mg) IV or
  * Cisplatin 75mg/m2 IV
  Interventions: Drug: Pegilodecakin; Drug: Paclitaxel or Docetaxel and Carboplatin or Cisplatin
- Part B: Dose Expansion Cohort (Experimental): Daily SC injection with pegilodecakin with Platinum / Taxane combination Every 21 days, (21 days = 1 cycle) for 5 cycles.
  Day 1
  * Paclitaxel 200/175 mg/m2 IV, or
  * Docetaxel 75/65 mg/m2 IV And
  * Carboplatin AUC 6/5/4 (max. 6x 150mg) IV or
  * Cisplatin 75mg/m2 IV
  Interventions: Drug: Pegilodecakin; Drug: Paclitaxel or Docetaxel and Carboplatin or Cisplatin
- Part C: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (2.5 ug/kg) daily subcutaneous injections with FOLFOX4 every 14 days FOLFOX4; (14 days = 1 cycle) ;
  Day 1
  * Oxaliplatin 85 mg/m2 IV over 2 hours
  * Leucovorin 200 mg/m2 IV over 2 hours followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  * Leucovorin 200 mg/m2 IV over 2 hours on Day 2 followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  Interventions: Drug: Pegilodecakin; Drug: FOLFOX (Oxaliplatin/Leucovorin/5-Fluorouracil)
- Part C: Dose Escalation Cohort 2 (Experimental): Pegilodecakin (5 ug/kg) daily subcutaneous injections with FOLFOX4 every 14 days FOLFOX4; (14 days = 1 cycle) ;
  Day 1
  * Oxaliplatin 85 mg/m2 IV over 2 hours
  * Leucovorin 200 mg/m2 IV over 2 hours followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  * Leucovorin 200 mg/m2 IV over 2 hours on Day 2 followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  Interventions: Drug: Pegilodecakin; Drug: FOLFOX (Oxaliplatin/Leucovorin/5-Fluorouracil)
- Part C: Dose Escalation Cohort 3 (Experimental): Pegilodecakin (10 ug/kg) daily subcutaneous injections with FOLFOX4 every 14 days FOLFOX4; (14 days = 1 cycle) ;
  Day 1
  * Oxaliplatin 85 mg/m2 IV over 2 hours
  * Leucovorin 200 mg/m2 IV over 2 hours followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  * Leucovorin 200 mg/m2 IV over 2 hours on Day 2 followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  Interventions: Drug: Pegilodecakin; Drug: FOLFOX (Oxaliplatin/Leucovorin/5-Fluorouracil)
- Part C: Dose Expansion Cohort 1 (Experimental): Daily SC injection with pegilodecakin with FOLFOX4 Every 14 days FOLFOX4; (14 days = 1 cycle) ;
  Day 1
  * Oxaliplatin 85 mg/m2 IV over 2 hours
  * Leucovorin 200 mg/m2 IV over 2 hours followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  * Leucovorin 200 mg/m2 IV over 2 hours on Day 2 followed by
  * 5-FU 400 mg/m2 IV bolus and
  * 5-FU 600 mg/m2/day IV over 22 hours
  Interventions: Drug: Pegilodecakin; Drug: FOLFOX (Oxaliplatin/Leucovorin/5-Fluorouracil)
- Part D: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (5 ug/kg) daily subcutaneous injections with Gemcitabine and nab-paclitaxel on Days 1, 8, 15 of each cycle (28 days = 1 cycle).
  Nab-paclitaxel 125 mg/m2 IV over 30 minutes followed by
  • Gemcitabine 1000 mg/m2 IV.
  Interventions: Drug: Pegilodecakin; Drug: gemcitabine/nab-paclitaxel
- Part E: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (10 ug/kg) daily subcutaneous injections with capecitabine BID daily for 14 days of each cycle (21 days= 1 cycle).
  • Capecitabine 1000 mg/m2 po BID
  Interventions: Drug: Pegilodecakin; Drug: Capecitabine
- Part F: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (10 ug/kg) daily subcutaneous injections with paclitaxel on Days 1, 8, 15 of each cycle (28 days= 1 cycle)
  • Paclitaxel 80 mg/ m2 IV
  Interventions: Drug: Pegilodecakin; Drug: Paclitaxel
- Part G: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (10 ug/kg) daily subcutaneous injections with pazopanib orally given daily for 14 days of each cycle (21 days= 1 cycle)
  • Pazopanib 800 mg po QD
  Interventions: Drug: Pegilodecakin; Drug: Pazopanib
- Part H: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (10 ug/kg) daily subcutaneous injections with pembrolizumab on Day 1 of each cycle (21 days= 1 cycle).
  • Pembrolizumab 2 mg/kg IV over 30 min
  Interventions: Drug: Pegilodecakin; Drug: Pembrolizumab
- Part I: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (20 ug/kg) daily subcutaneous injections with nivolumab on Day 1 of each cycle (14 days= 1 cycle).
  • Nivolumab 3 mg/kg IV over 60 min
  Interventions: Drug: nivolumab
- Part H: Dose Escalation Cohort 2 (Experimental): Pegilodecakin (20 ug/kg) daily subcutaneous injections with pembrolizumab on Day 1 of each cycle (21 days= 1 cycle).
  • Pembrolizumab 2 mg/kg IV over 30 min
  Interventions: Drug: Pembrolizumab
- Part H: Dose Escalation Cohort 3 (Experimental): Pegilodecakin (40 ug/kg) daily subcutaneous injections with pembrolizumab on Day 1 of each cycle (21 days= 1 cycle).
  • Pembrolizumab 2 mg/kg IV over 30 min
  Interventions: Drug: Pembrolizumab
- Part J: Dose Escalation Cohort 1 (Experimental): Pegilodecakin (10 ug/kg) daily subcutaneous injections with gemcitabine and carbolplatin on Days 1,8 of each cycle (21 days=1 cycle) until disease progression gemcitabine 1000mg/m2 IV over 30 minutes followed by carboplatin AUC2 over 60 minutes
  Interventions: Drug: Gemcitabine/carboplatin

INTERVENTIONS:
Drug: Pegilodecakin — Daily subcutaneous injections of pegilodecakin up to 12 months
  Other Names: LY3500518; AM0010; PEGylated recombinant human Interleukin-10; PEG-rHuIL-10
  Arms: Part A: Dose Escalation Cohort 1; Part A: Dose Escalation Cohort 2; Part A: Dose Escalation Cohort 3; Part A: Dose Escalation Cohort 4; Part A: Dose Escalation Cohort 5; Part A: Dose Escalation Cohort 6; Part A: Dose Expansion Cohort 1; Part B: Dose Escalation Cohort 1; Part B: Dose Escalation Cohort 2; Part B: Dose Escalation Cohort 3; Part B: Dose Expansion Cohort; Part C: Dose Escalation Cohort 1; Part C: Dose Escalation Cohort 2; Part C: Dose Escalation Cohort 3; Part C: Dose Expansion Cohort 1; Part D: Dose Escalation Cohort 1; Part E: Dose Escalation Cohort 1; Part F: Dose Escalation Cohort 1; Part G: Dose Escalation Cohort 1; Part H: Dose Escalation Cohort 1
Drug: Paclitaxel or Docetaxel and Carboplatin or Cisplatin — Day 1 of every 21 day cycle
  Other Names: Taxol or taxotere and paraplatin or platinol
  Arms: Part B: Dose Escalation Cohort 1; Part B: Dose Escalation Cohort 2; Part B: Dose Escalation Cohort 3; Part B: Dose Expansion Cohort
Drug: FOLFOX (Oxaliplatin/Leucovorin/5-Fluorouracil) — Intravenous administration on Day 1 and 2 of every 14 day cycle
  Other Names: Eloxatin®/Leucovorin/5-FU
  Arms: Part C: Dose Escalation Cohort 1; Part C: Dose Escalation Cohort 2; Part C: Dose Escalation Cohort 3; Part C: Dose Expansion Cohort 1
Drug: gemcitabine/nab-paclitaxel — Intravenous administration of the gemcitabine/nab-paclitaxel regimen on Day 1, 8 and 15 of each 28 day treatment cycle.
  Other Names: Gemzar/Abraxane ABI-007
  Arms: Part D: Dose Escalation Cohort 1
Drug: Capecitabine — Capecitabine will be administered orally twice daily for 14 days out of every 21 days.
  Other Names: Xeloda
  Arms: Part E: Dose Escalation Cohort 1
Drug: Pazopanib — Pazopanib will be administered orally daily continuously
  Other Names: GW786034
  Arms: Part G: Dose Escalation Cohort 1
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously on Day 1 of every 21 day cycle.
  Other Names: Keytruda, MK-3475
  Arms: Part H: Dose Escalation Cohort 1; Part H: Dose Escalation Cohort 2; Part H: Dose Escalation Cohort 3
Drug: Paclitaxel — Paclitaxel will be administered intravenously on Days 1, 8, 15 of each cycle (28 days= 1 cycle)
  • Paclitaxel 80 mg/ m2 IV
  Arms: Part F: Dose Escalation Cohort 1
Drug: nivolumab — Nivolumab on Day 1 of each cycle (14 days = 1 cycle)
  Other Names: Keytruda
  Arms: Part I: Dose Escalation Cohort 1
Drug: Gemcitabine/carboplatin — gemcitabine and carboplatin on Days 1, 8 of each cycle (21 days = 1 cycle)
  Other Names: gemzar/paraplatin
  Arms: Part J: Dose Escalation Cohort 1

SUMMARY:
This is a first-in-human, open-label, dose escalation study to evaluate the safety and tolerability of pegilodecakin in participants with advanced solid tumors, dosed daily subcutaneously as a monotherapy or in combination with chemotherapy or immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Part A Escalation Cohorts:

o Histologically or cytologically confirmed advanced malignant solid tumor, limited to melanoma, castrate resistant prostate cancer (CRPC), ovarian cancer (OVCA), renal cell carcinoma, colorectal carcinoma (CRC), pancreatic carcinoma or non-small cell lung carcinoma (NSCLC) that is refractory to, intolerant of, for which no standard of therapy is available or where the participant refuses existing therapies

Part A Expansion Cohorts, Part B and C Escalation and Expansion Cohorts:

* Tumors with all histological diagnosis or tissue origin may be enrolled
* Participants must have failed prior standard curative chemotherapy for their disease, refuse existing therapies OR the proposed chemotherapy regimen to which pegilodecakin is added represents an acceptable standard treatment for their disease.

  * Measurable or evaluable disease according to irRC or bone metastatic disease evaluable by Prostate Cancer Working Group 2 criteria (PCWG2) for castration-resistant prostate cancer (CRPC)
  * At least 18 years of age
  * Performance Status of 0 or 1
  * Adequate organ function

Exclusion Criteria:

* Hematologic malignancies
* Pregnant or lactating
* Present or history of neurological disorders such as Multiple Sclerosis and Guillain Barre or inflammatory central nervous system/peripheral nervous system (CNS/PNS) disorders
* Myocardial infarction within the last 6 months
* Unstable angina, or unstable cardiac arrhythmia requiring medication
* Surgery within the last 28 days
* Systemic fungal, bacterial, viral, or other infection
* History of bleeding diathesis within the last 6 months
* Positive for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2013-11-15 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as measured by incidence of adverse events | up to 12 months
Pharmacokinetic (PK) parameters | up to 12 months
  PK parameters including the serum trough concentration (Minimal Drug Concentration (Cmin)), the maximal drug concentration (Cmax), area under the curve of serum concentration over time (Area Under the Curve/ AUC), and half-life (t½).

SECONDARY OUTCOMES:
Change in tumor burden measured by volumetric Computer Tomography (CT) or Magnetic Resonance Imaging (MRI) according to immune-related response criteria (irRC) | up to 12 months
Progression in bone by bone scintigraphy according to Prostate Cancer Working Group 2 (PCWG2) for participants with metastatic castration resistant prostate cancer (CRPC) | approximatley 4 months
Anti-Pegilodecakin antibody formation | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - UCLA Medical Hematology & Oncology, Los Angeles, California
  - UCSF, San Francisco, California
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stephenson Cancer Center at Oklahoma University TSET Phase 1 Program, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naing A, Wong DJ, Infante JR, Korn WM, Aljumaily R, Papadopoulos KP, Autio KA, Pant S, Bauer TM, Drakaki A, Daver NG, Hung A, Ratti N, McCauley S, Van Vlasselaer P, Verma R, Ferry D, Oft M, Diab A, Garon EB, Tannir NM. Pegilodecakin combined with pembrolizumab or nivolumab for patients with advanced solid tumours (IVY): a multicentre, multicohort, open-label, phase 1b trial. Lancet Oncol. 2019 Nov;20(11):1544-1555. doi: 10.1016/S1470-2045(19)30514-5. Epub 2019 Sep 25. PMID 31563517
- [Derived] Naing A, Papadopoulos KP, Autio KA, Ott PA, Patel MR, Wong DJ, Falchook GS, Pant S, Whiteside M, Rasco DR, Mumm JB, Chan IH, Bendell JC, Bauer TM, Colen RR, Hong DS, Van Vlasselaer P, Tannir NM, Oft M, Infante JR. Safety, Antitumor Activity, and Immune Activation of Pegylated Recombinant Human Interleukin-10 (AM0010) in Patients With Advanced Solid Tumors. J Clin Oncol. 2016 Oct 10;34(29):3562-3569. doi: 10.1200/JCO.2016.68.1106. PMID 27528724